CLINICAL TRIAL: NCT06930508
Title: Implementing HIV Pre-Exposure Prophylaxis in a Family Planning Clinic: A Study of Feasibility and Acceptability (Aka The Pilot Fish Study)
Brief Title: Bringing Medicines for HIV Prevention to a Family Planning Clinic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Advance RI CTR (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2282543-1
Record Dates: First submitted 2025-04-01; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: HIV; PrEP
Keywords: HIV PrEP screening; HIV PrEP initiation; ob/gyn

STUDY DESIGN:
Intervention Model Description: There will be no between-group comparison in this trial. However, the investigators will simultaneously recruit both patient participants and physician participants. Study procedures will be different for these two groups, as described in the protocol section.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Participant (Experimental)
  Interventions: Behavioral: Patient participant screening
- Physician Participant (Experimental)
  Interventions: Behavioral: Physician participant training

INTERVENTIONS:
Behavioral: Patient participant screening — Patient participants will be provided with the standardized PrEP screening and initiation protocol.
  Arms: Patient Participant
Behavioral: Physician participant training — Physician participants will be trained in the investigators' standardized PrEP screening and initiation protocol.
  Arms: Physician Participant

SUMMARY:
The goal of this clinical trial is to understand what patients and physicians think about providing medications to prevent HIV transmission to patients in a family planning clinic. These medications are known as pre-exposure prophylaxis, or PrEP. The main questions to answer are:

1. Do patients find it acceptable to be asked about, and offered, PrEP during their visit to a family planning clinic?
2. What things make it easier or harder to ask about PrEP in a family planning clinic setting?
3. What things make it easier or harder to begin PrEP in a family planning clinic setting?

Patient participants:

1. Will receive standardized counseling about PrEP.
2. Will have the opportunity to begin PrEP as part of their routine, ongoing care.
3. Will be asked to complete a survey about their experiences.

Physician participants:

1. Will receive standardized education about PrEP.
2. Will talk to patient participants about PrEP, and support patient participants who want to begin PrEP.
3. Will be asked to complete pre-and post-study surveys about their experiences.
4. May be asked to complete a post-study in-depth interview about their experiences.

DETAILED DESCRIPTION:
In the proposed pilot study, the investigators' goal is to improve community health resources available to Rhode Islanders to lower their risk of HIV acquisition, via the following specific aims:

1. Evaluate the patient acceptability of HIV pre-exposure prophylaxis (PrEP) eligibility screening and initiation in an ob/gyn-staffed family planning clinic.
2. Assess the barriers, facilitators, and feasibility of PrEP eligibility screening in an ob/gyn-staffed family planning clinic.
3. Assess the barriers, facilitators, and feasibility of delivery and uptake of PrEP in an ob/gyn-staffed family planning clinic.

Overall, the investigators' expected outcome is to have exploratory data to inform a scalable intervention to implement PrEP access, which can be deployed in family planning clinic settings, and which is designed in accordance with acceptability and feasibility data from patients and providers. Since the existing data suggest that ob/gyn-staffed family planning clinics are an ideal site both as a catchment area for patients who are at higher risk for HIV acquisition, and in terms of technical capacity and provider skill set, the next step to expand PrEP service delivery in these settings is to assess the barriers and facilitators to such care, in order to meet patients where they are, with the care they need. The goal is to situate the protocol to fit into the usual clinical workflow of a busy family planning clinic.

The investigators will develop and implement a standardized PrEP eligibility screening instrument and initiation protocol, based on CDC guidelines. The investigators will survey patient and physician participants about feasibility and acceptability of study procedures. Patient participants will be approached by a research assistant, who will inform eligible individuals about the purpose, risks, and benefits of the study. The research assistant will obtain informed consent from participants. Physicians will then screen participants for PrEP eligibility per protocol, and will offer initiation of PrEP. These medications are not investigational, are part of standard of care STI prevention, and are not themselves the primary subject of this study.

The investigators' primary data collection will be via survey. Patient participants will receive a $25 gift card for completing the post-intervention survey. Physician participants will receive pre- and post-study surveys, and a subgroup will participate in focused interviews.

There is no control arm in this study. The alternative to participation in this study is to simply undergo (or provide) routine care in the investigators' Family Planning Clinic, which does not currently include PrEP provision - though, as described above, such care is within the scope of routine care in ob/gyn settings.

ELIGIBILITY:
This study will include patient participants who:

* Are age 16 or older
* Are presenting for care at the Women and Infants Hospital of Rhode Island Family Planning Clinic
* Speak English or Spanish
* Have decisional capacity

This study will exclude patient participants who:

- Are currently seeking abortion care

This study will include physician participants who:

- Provide care at the Women and Infants Hospital of Rhode Island Family Planning Clinic

This study will not have any specific exclusion criteria for physician participants.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Post-visit questionnaire | Once, at the end of the study visit
  Patient participants will receive post-visit questionnaires to assess Specific Aims 1, 2, and 3.
Pre- and post-study questionnaires | Once, at study enrollment, and once at the completion of physician participation in the study (maximum anticipated timeframe, 1 year)
  Physician participants will receive pre- and post-study questionnaires to assess Specific Aims 2 and 3.

SECONDARY OUTCOMES:
Qualitative interviews | Once at the completion of physician participation in the study (maximum anticipated timeframe, 1 year)
  A subgroup of physician participants will be engaged in qualitative interviews to further contextualize their survey responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Women and Infants Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No